CLINICAL TRIAL: NCT00844285
Title: A Non-Interventional Long-term Post-Marketing Registry of Patients Treated With Certolizumab Pegol (Cimzia ®) for Crohn's Disease
Brief Title: SECURE, the Cimzia ® Crohn's Disease Post-Marketing Registry
Acronym: SECURE
Status: Completed | Type: Observational
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: C87075
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Crohn's Disease
Keywords: Certolizumab Pegol, Cimzia ®; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cimzia Cohort:: Patients about to receive treatment with Cimzia® as part of pre-existing management plan for Crohn's disease or has already been receiving treatment with Cimzia® for ≤12 months. Patients must also receive a Cimzia dose within 2 months following enrollment.
  Interventions: Drug: Cimzia
- Comparison cohort: Patient must be about to receive treatment with any other medication as part of a pre-existing management plan for Crohn's disease or has already been receiving treatment (previous Cimzia® treatment is prohibited).

INTERVENTIONS:
Drug: Cimzia — The associated drug description is a total of two 200 mg subcutaneous injections of Cimzia to total 400 mg.
  Groups: Cimzia Cohort:

SUMMARY:
The purpose of this study is to monitor safety outcomes of patients who have taken Cimzia® as compared to a non- Cimzia® control population. The SECURE Registry's target enrollment is 3045 patients and it's objective is to monitor patients for approximately 8 years.

DETAILED DESCRIPTION:
Physicians are expected to manage patients as they would under normal practice conditions; patients will receive and use their medications according to their normal course of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have medically documented Crohn's disease (CD)
* The decision to prescribe Cimzia or other medications has been made by the physician independent of inclusion in this study
* Patient (or his/her legally acceptable representative) is able to provide written informed consent to permit collection of data
* Patients participating in randomized, blinded clinical trials for CD or other conditions are not eligible for inclusion into the SECURE registry. Involvement in other registries, where patients follow routine clinical practice, is permitted, however
* For the Cimzia cohort: Patient is receiving treatment with Cimzia for the first time. Patient must receive Cimzia treatment within 2 months of enrollment into the registry
* Patient is currently receiving treatment with Cimzia for <=12 months. Patient must also receive a Cimzia dose within 2 months following enrollment into the registry
* For the comparison cohort: Patient is switching CD treatment or beginning CD treatment for the first time. Previous Cimzia treatment is prohibited in the comparator group. Patient must receive new CD treatment within 2 months of enrollment into the registry. Patient is currently receiving anti-TNF treatment for <=12 months. Patient must receive anti-TNF treatment within 2 months following enrollment into the registry. Patient is currently receiving immunosuppressant therapy for <=12 months. Patient must receive immunosuppressant therapy within 2 months following enrollment into the registry. Patient is currently receiving systemic steroid therapy for <=12 months. Patient must receive systemic steroid therapy within 2 months following enrollment into registry.

Exclusion Criteria:

* See inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of selected gastroenterologists and internal medicine physicians from both community-based and academic practice settings (75% and 25% respectively) Each physician should be able to recruit a minimum of 5 patients prescribed Cimzia® and/or 5 patients prescribed other treatments.
  Recruitment into both cohorts will be monitored and controlled as needed in order to ensure balanced enrollment over time. In order to ensure reasonable balance between both cohorts, retrospective frequency matching will be applied for disease severity (mild/moderate/severe), age categories and gender.
Sampling Method: Non-Probability Sample
Enrollment: 3072 (Actual)
Dates: Start 2009-01-30 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273(UCB)
Locations (197):
- United States (197):
  - C87075 931, Birmingham, Alabama
  - C87075 198, Birmingham, Alabama
  - C87075 286, Huntsville, Alabama
  - C87075 032, Montgomery, Alabama
  - C87075 253, Scottsdale, Arizona
  - C87075 307, Tucson, Arizona
  - C87075 377, Tucson, Arizona
  - C87075 574, North Little Rock, Arkansas
  - C87075 059, Beverly Hills, California
  - C87075 580, Encino, California
  - C87075 021, Fountain Valley, California
  - C87075 261, La Jolla, California
  - C87075 220, Los Angeles, California
  - C87075 728, Oceanside, California
  - C87075 571, Palm Springs, California
  - C87075 485, San Carlos, California
  - C87075 027, Torrance, California
  - C87075 946, Boulder, Colorado
  - C87075 491, Lonetree, Colorado
  - C87075 087, Hamden, Connecticut
  - C87075 077, Hartford, Connecticut
  - C87075 097, Torrington, Connecticut
  - C87075 639, Altamonte Springs, Florida
  - C87075 049, Boca Raton, Florida
  - C87075 871, Boca Raton, Florida
  - C87075 002, Gainesville, Florida
  - C87075 759, Hialeah, Florida
  - C87075 893, Hollywood, Florida
  - C87075 143, Lakeland, Florida
  - C87075 970, Largo, Florida
  - C87075 030, Lauderdale Lakes, Florida
  - C87075 009, Maitland, Florida
  - C87075 003, Miami, Florida
  - C87075 004, Miami, Florida
  - C87075 102, Miami, Florida
  - C87075 420, Miami, Florida
  - C87075 034, Naples, Florida
  - C87075 031, Orlando, Florida
  - C87075 487, Orlando, Florida
  - C87075 935, Orlando, Florida
  - C87075 074, Palm Coast, Florida
  - C87075 183, Sarasota, Florida
  - C87075 144, Tampa, Florida
  - C87075 046, Titusville, Florida
  - C87075 271, Vero Beach, Florida
  - C87075 280, Weston, Florida
  - C87075 729, Winter Park, Florida
  - C87075 399, Atlanta, Georgia
  - C87075 288, Atlanta, Georgia
  - C87075 849, Atlanta, Georgia
  - C87075 232, Covington, Georgia
  - C87075 357, Cumming, Georgia
  - C87075 336, Decatur, Georgia
  - C87075 113, Decatur, Georgia
  - C87075 988, Decatur, Georgia
  - C87075 698, Johns Creek, Georgia
  - C87075 083, Lawrenceville, Georgia
  - C87075 067, Macon, Georgia
  - C87075 897, Macon, Georgia
  - C87075 488, Marietta, Georgia
  - C87075 229, Boise, Idaho
  - C87075 245, Idaho Falls, Idaho
  - C87075 037, Meridian, Idaho
  - C87075 278, Arlington Heights, Illinois
  - C87075 418, Chicago, Illinois
  - C87075 168, Chicago, Illinois
  - C87075 858, Evanston, Illinois
  - C87075 208, Hoffman Estates, Illinois
  - C87075 368, Oak Lawn, Illinois
  - C87075 370, Oakbrook Terrace, Illinois
  - C87075 151, Indianapolis, Indiana
  - C87075 124, Indianapolis, Indiana
  - C87075 343, Clive, Iowa
  - C87075 204, Lexington, Kentucky
  - C87075 072, Baton Rouge, Louisiana
  - C87075 214, Hammond, Louisiana
  - C87075 108, Metairie, Louisiana
  - C87075 997, New Orleans, Louisiana
  - C87075 987, Shreveport, Louisiana
  - C87075 235, Annapolis, Maryland
  - C87075 040, Annapolis, Maryland
  - C87075 181, Baltimore, Maryland
  - C87075 953, Baltimore, Maryland
  - C87075 591, Towson, Maryland
  - C87075 091, Boston, Massachusetts
  - C87075 567, Boston, Massachusetts
  - C87075 395, Newton, Massachusetts
  - C87075 939, North Adams, Massachusetts
  - C87075 869, Ann Arbor, Michigan
  - C87075 260, Chesterfield, Michigan
  - C87075 195, Kalamazoo, Michigan
  - C87075 349, Novi, Michigan
  - C87075 579, Troy, Michigan
  - C87075 373, Wyandotte, Michigan
  - C87075 167, Wyoming, Michigan
  - C87075 843, Wyoming, Michigan
  - C87075 829, Ypsilanti, Michigan
  - C87075 215, Plymouth, Minnesota
  - C87075 501, Rochester, Minnesota
  - C87075 867, Ocean Springs, Mississippi
  - C87075 540, Bridgeton, Missouri
  - C87075 163, Columbia, Missouri
  - C87075 776, Lee's Summit, Missouri
  - C87075 305, Mexico, Missouri
  - C87075 085, St Louis, Missouri
  - C87075 835, St Louis, Missouri
  - C87075 937, Las Vegas, Nevada
  - C87075 740, Lebanon, New Hampshire
  - C87075 323, Nashua, New Hampshire
  - C87075 005, Cherry Hill, New Jersey
  - C87075 705, Egg Harbor, New Jersey
  - C87075 930, Marlton, New Jersey
  - C87075 610, Mays Landing, New Jersey
  - C87075 161, Ridgewood, New Jersey
  - C87075 165, Woodbury, New Jersey
  - C87075 024, Brooklyn, New York
  - C87075 362, Flushing, New York
  - C87075 413, Great Neck, New York
  - C87075 517, Great Neck, New York
  - C87075 321, Jericho, New York
  - C87075 541, Lake Success, New York
  - C87075 118, New York, New York
  - C87075 712, New York, New York
  - C87075 494, New York, New York
  - C87075 018, New York, New York
  - C87075 159, Poughkeepsie, New York
  - C87075 300, Rochester, New York
  - C87075 884, Stony Brook, New York
  - C87075 051, Asheville, North Carolina
  - C87075 636, Chapel Hill, North Carolina
  - C87075 185, Charlotte, North Carolina
  - C87075 965, Charlotte, North Carolina
  - C87075 945, Concord, North Carolina
  - C87075 973, Fayetteville, North Carolina
  - C87075 527, Greenville, North Carolina
  - C87075 127, Kinston, North Carolina
  - C87075 926, New Bern, North Carolina
  - C87075 779, Rocky Mount, North Carolina
  - C87075 932, Wilmington, North Carolina
  - C87075 955, Bismarck, North Dakota
  - C87075 239, Canton, Ohio
  - C87075 807, Canton, Ohio
  - C87075 042, Cincinnati, Ohio
  - C87075 016, Cincinnati, Ohio
  - C87075 462, Cleveland, Ohio
  - C87075 314, Lima, Ohio
  - C87075 929, Mentor, Ohio
  - C87075 777, Tulsa, Oklahoma
  - C87075 172, Tulsa, Oklahoma
  - C87075 213, Portland, Oregon
  - C87075 947, Allentown, Pennsylvania
  - C87075 241, Hermitage, Pennsylvania
  - C87075 460, Malvern, Pennsylvania
  - C87075 166, Philadelphia, Pennsylvania
  - C87075 086, Pittsburgh, Pennsylvania
  - C87075 176, Charleston, South Carolina
  - C87075 813, Columbia, South Carolina
  - C87075 922, Sioux Falls, South Dakota
  - C87075 299, Franklin, Tennessee
  - C87075 262, Hermitage, Tennessee
  - C87075 757, Jackson, Tennessee
  - C87075 224, Knoxville, Tennessee
  - C87075 390, Nashville, Tennessee
  - C87075 894, Nashville, Tennessee
  - C87075 596, Union City, Tennessee
  - C87075 272, Austin, Texas
  - C87075 200, Austin, Texas
  - C87075 941, Dallas, Texas
  - C87075 628, Dallas, Texas
  - C87075 088, Fort Sam Houston, Texas
  - C87075 226, Fort Worth, Texas
  - C87075 237, Houston, Texas
  - C87075 419, Houston, Texas
  - C87075 726, Houston, Texas
  - C87075 312, Pasadena, Texas
  - C87075 657, San Antonio, Texas
  - C87075 923, San Antonio, Texas
  - C87075 279, Southlake, Texas
  - C87075 366, Temple, Texas
  - C87075 539, Tyler, Texas
  - C87075 986, Salt Lake City, Utah
  - C87075 814, Burlington, Vermont
  - C87075 963, Colchester, Vermont
  - C87075 675, Christiansburg, Virginia
  - C87075 691, Norfolk, Virginia
  - C87075 446, Richmond, Virginia
  - C87075 026, Virginia Beach, Virginia
  - C87075 273, Woodbridge, Virginia
  - C87075 471, Seattle, Washington
  - C87075 925, Tacoma, Washington
  - C87075 465, Green Bay, Wisconsin
  - C87075 116, Madison, Wisconsin
  - C87075 070, Milwaukee, Wisconsin
  - C87075 281, Milwaukee, Wisconsin
  - C87075 389, Milwaukee, Wisconsin
  - C87075 578, Milwaukee, Wisconsin
  - C87075 093, Oshkosh, Wisconsin

REFERENCES:
- [Derived] Lichtenstein GR, Lee SD, Feagan BG, Loftus EV Jr, Ng S, Dehlin K, Quinn P, Coarse J, Rosario-Jansen T, Arendt C, Stark JL. Certolizumab Pegol Treatment in Patients With Crohn's Disease: Final Safety Data From the SECURE Registry. Crohns Colitis 360. 2025 Jan 25;7(1):otae083. doi: 10.1093/crocol/otae083. eCollection 2025 Jan. PMID 39895830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in January 2009 and concluded in August 2020.
Pre-assignment Details: Participant flow refers to the Enrolled Set.
Groups:
- Cimzia at Baseline: Participants who received Cimzia® up to 70 days prior to Baseline.
- No Cimzia at Baseline: Participants not in the Cimzia® at Baseline group receiving corticosteroids, immunosuppressants or other biologics (e.g. anti-TNFs) other than Cimzia® at Baseline.
- Gap (No Cimzia and no Comparator at Baseline): Participants who did not receive Cimzia® within 70 days prior to Baseline nor corticosteroids, immunosuppressants or other biologics (e.g. anti-TNFs) other than Cimzia® at Baseline.
Period: Overall Study
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline)
Started | 1131 | 1666 | 275
Completed | 42 | 62 | 3
Not Completed | 1089 | 1604 | 272
Not completed — Other | 0 | 1 | 0
Not completed — Other than specified | 95 | 129 | 12
Not completed — Site closure | 256 | 450 | 50
Not completed — Follow-up < 8 years | 16 | 23 | 4
Not completed — Protocol Violation | 26 | 28 | 54
Not completed — Death | 22 | 21 | 8
Not completed — Withdrew Consent | 344 | 466 | 70
Not completed — Lost to Follow-up | 330 | 486 | 74

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Enrolled Set which was defined as all participants enrolled and with an informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline) | Total
Number analyzed (Participants) | 1131 | 1666 | 275 | 3072
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 71 | 10 | 115
  Between 18 and 65 years | 1018 | 1510 | 222 | 2750
  >=65 years | 79 | 85 | 43 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (14.9) | 39.2 (14.9) | 45.0 (17.8) | 40.0 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 706 | 924 | 166 | 1796
  Male | 425 | 740 | 104 | 1269
  Missing | 0 | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian /Alaskan native | 2 | 4 | 1 | 7
  Asian | 13 | 19 | 3 | 35
  Black | 82 | 117 | 13 | 212
  Native Hawaiian or other Pacific Islander | 1 | 2 | 4 | 7
  White | 1017 | 1480 | 243 | 2740
  Other/mixed | 14 | 35 | 5 | 54
  Missing | 2 | 9 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 79 | 19 | 142
  Not Hispanic or Latino | 1086 | 1585 | 250 | 2921
  Missing | 1 | 2 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events of Interest Per 100 Participants-Years By Actual Treatment (Malignancy Rules)
Description: Incidence rate is defined as the number of participants experiencing the event of interest divided by the number person-years without an event (time up to the event for participants experiencing an event, and the full study time for those without). Adverse events of interest included malignant or unspecified tumor, serious infections, opportunistic infections, serious cardiovascular events, congestive heart failure, demyelinating-like disorders, aplastic anemia, pancytopenia, thrombocytopenia, neutropenia, leucopenia, serious bleeding events, lupus and lupus-like illness, serious skin reactions, hepatic events, hypersensitivity reactions and anaphylactic reactions, malignant lymphomas, non-melanoma skin cancer, autoimmune disorders. Treatment groups are based upon actual treatment conservatively assigning participant time and events to CZP even after stopping CZP. Data for malignant or unspecified tumor as per malignancy rules has been reported in this outcome measure.
Time Frame: Baseline up to 10 years
Population: Enrolled set was defined as all participants enrolled and with an informed consent. Here, "Number of Participants Analyzed" included those who were evaluable for this outcome measure. Participants were counted in more than one arm based on the various treatments they actually received and presented. Based upon planned analysis, data is reported for Cimzia® and Comparator reporting groups only.
Measure: Number (95% Confidence Interval); unit: no. of events per 100 participant-years
Groups:
- Cimzia: Participants (exposure and events) are conservatively included in this group from the time of first administration of Cimzia® until the end of the study even if they switch to comparator. Participants may be included in other treatment groups.
- Comparator: Participants (exposure and events) are included in this group from the time of first administration of comparator until the end of the study or switch to Cimzia®, a participant cannot be in the comparator group if their first treatment in the study was Cimzia®. Participants may be included in other treatment groups.
Arm/Group | Cimzia | Comparator
Number analyzed (Participants) | 1463 | 1887
no. of events per 100 participant-years | 0.45 [0.31 to 0.65] | 0.65 [0.48 to 0.86]

2. Primary Outcome: Incidence of Adverse Events of Interest Per 100 Participant-Years By Actual Treatment (Acute Event Rules)
Description: Incidence rate is defined as the number of participants experiencing the event of interest divided by the number person-years without an event (time up to the event for participants experiencing an event, and the full study time for those without an event of interest). Adverse events of interest (AEoI) included malignant or unspecified tumor, serious infections, opportunistic infections, serious cardiovascular events, congestive heart failure, demyelinating-like disorders, aplastic anemia, pancytopenia, thrombocytopenia, neutropenia, leucopenia, serious bleeding events, lupus and lupus-like illness, serious skin reactions, hepatic events, hypersensitivity reactions and anaphylactic reactions, malignant lymphomas, non-melanoma skin cancer, autoimmune disorders. Data for AEoIs as per acute event rules has been reported in this outcome measure where the AEoI is assigned to the treatment the participant is on at the time of the event.
Time Frame: Baseline up to 10 years
Population: Enrolled set was defined as all participants enrolled and with an informed consent. Here, "Number of Participants Analyzed" included those who were evaluable for this outcome measure. Participants were counted in more than one arm based on the various treatments they actually received and presented. Based upon planned analysis, data is reported for Cimzia®, Comparator, Overlap, Gap and Cimzia®+Overlap reporting groups only.
Measure: Number (95% Confidence Interval); unit: no. of events per 100 participant-years
Groups:
- Cimzia: Participants (exposure and events) while receiving Cimzia® alone, including the half-life of Cimzia® unless comparator is started during this time. Participants may be included in other treatment groups.
- Comparator: Participants (exposure and events) while receiving corticosteroids, immunosuppressants or other biologics (e.g. anti-TNFs) other than Cimzia®, alone or in combination with each other including their half-life. Participants may be included in other treatment groups.
- Overlap: Participants (exposure and events) while receiving Cimzia® along with corticosteroids, immunosuppressants or other biologics (e.g. anti-TNFs) other than Cimzia® including the half-life time of Cimzia® and the comparator. Participants may be included in other treatment groups.
- Gap (No Cimzia and no Comparator at Baseline): Participants (exposure and events) neither receiving Cimzia® (including the half-life of Cimzia®) nor receiving comparator (including the half-life). Participants may be included in other treatment groups.
- Cimzia + Overlap: Participants who received Cimzia® monotherapy or Cimzia® in combination with comparison treatment were included in this group. Participants may be included in other treatment groups.
Arm/Group | Cimzia | Comparator | Overlap | Gap (No Cimzia and no Comparator at Baseline) | Cimzia + Overlap
Number analyzed (Participants) | 824 | 2478 | 1165 | 1022 | 1428
no. of events per 100 participant-years
  Malignant or Unspecified Tumor | 0.35 [0.12 to 0.83] | 0.59 [0.44 to 0.77] | 0.60 [0.28 to 1.15] | 0.56 [0.29 to 0.97] | 0.48 [0.26 to 0.81]
  Serious infections | 2.03 [1.35 to 2.94] | 1.59 [1.34 to 1.88] | 6.15 [4.90 to 7.61] | 1.46 [0.98 to 2.08] | 4.08 [3.36 to 4.91]
  Opportunistic infections | 0.14 [0.02 to 0.50] | 0.08 [0.03 to 0.16] | 0.20 [0.04 to 0.59] | 0.09 [0.01 to 0.33] | 0.17 [0.06 to 0.40]
  Serious cardiovascular events | 0.14 [0.02 to 0.50] | 0.13 [0.07 to 0.23] | 0.34 [0.11 to 0.78] | 0.23 [0.07 to 0.53] | 0.24 [0.10 to 0.49]
  Congestive heart failure | 0 [0 to 0] | 0.08 [0.03 to 0.15] | 0.07 [0.00 to 0.37] | 0 [0 to 0] | 0.03 [0.00 to 0.19]
  Demyelinating-like disorders | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Aplastic Anemia, Pancytopenia, Thrombocytopenia, Neutropenia, Leucopenia | 0 [0 to 0] | 0.08 [0.03 to 0.15] | 0.27 [0.07 to 0.68] | 0.14 [0.03 to 0.40] | 0.14 [0.04 to 0.35]
  Serious bleeding events | 0.28 [0.08 to 0.73] | 0.23 [0.14 to 0.35] | 0.47 [0.19 to 0.97] | 0.14 [0.03 to 0.40] | 0.38 [0.19 to 0.68]
  Lupus and lupus-like illness | 0 [0 to 0] | 0.06 [0.02 to 0.14] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Serious skin reactions | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Hepatic Events | 0.07 [0.00 to 0.39] | 0.09 [0.04 to 0.17] | 0.13 [0.02 to 0.48] | 0.05 [0.00 to 0.25] | 0.10 [0.02 to 0.30]
  Hypersensitivity reactions and anaphylactic reactions | 0.28 [0.08 to 0.72] | 0.11 [0.05 to 0.20] | 0.60 [0.28 to 1.14] | 0 [0 to 0] | 0.44 [0.24 to 0.76]
  Malignant lymphomas | 0.07 [0.00 to 0.39] | 0.04 [0.01 to 0.11] | 0.13 [0.02 to 0.48] | 0 [0 to 0] | 0.10 [0.02 to 0.30]
  Non-melanoma skin cancer | 0.14 [0.02 to 0.51] | 0.24 [0.15 to 0.36] | 0.20 [0.04 to 0.59] | 0.05 [0.00 to 0.25] | 0.17 [0.06 to 0.40]
  Autoimmune disorders | 0.35 [0.11 to 0.82] | 0.36 [0.25 to 0.50] | 0.27 [0.07 to 0.69] | 0.23 [0.07 to 0.53] | 0.31 [0.14 to 0.59]

3. Secondary Outcome: Change From Baseline in Physician's Harvey Bradshaw Index (HBI) Total Score to Each Post-Baseline Assessment
Description: HBI measured 5 parameters: the general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), presence of an abdominal mass on physical exam (0= none to 3= definite and tender), and whether there are any complications [1 per item: joint pain (arthralgia), eye inflammation (uveitis), red nodules on skin (erythema nodosum), canker sores (aphthous ulcers), skin wound/ulcers (pyoderma gangrenosum), tear in skin of anal area (anal fissure), fluid or pus drainage from anal area (new fistula), and abscess]. The total HBI score was sum of all the 5 individual parameters, where minimum score was 0 and there was no pre-specified maximum score as it was dependent on the number of liquids stools. Higher HBI scores indicated greater disease activity. A negative change indicated less disease activity.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102, and 108, compared to Baseline
Population: Enrolled Set was defined as all participants enrolled and with an informed consent. Here, "Number Analyzed" included those who were evaluable at specified time points only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline)
Number analyzed (Participants) | 1131 | 1666 | 275
units on a scale
  Month 6: number analyzed (Participants) | 746 | 1009 | 156
  Month 6 | -1.1 (4.3) | -0.7 (3.8) | -1.3 (4.7)
  Month 12: number analyzed (Participants) | 596 | 893 | 135
  Month 12 | -1.2 (5.3) | -0.8 (3.8) | -1.3 (4.9)
  Month 18: number analyzed (Participants) | 491 | 794 | 120
  Month 18 | -1.6 (4.6) | -0.8 (4.2) | -1.8 (5.5)
  Month 24: number analyzed (Participants) | 429 | 723 | 111
  Month 24 | -1.9 (4.7) | -1.2 (3.7) | -1.3 (4.9)
  Month 30: number analyzed (Participants) | 361 | 630 | 97
  Month 30 | -1.6 (4.7) | -1.1 (3.9) | -1.1 (4.5)
  Month 36: number analyzed (Participants) | 328 | 573 | 90
  Month 36 | -1.8 (5.2) | -1.1 (3.6) | -1.9 (5.1)
  Month 42: number analyzed (Participants) | 291 | 501 | 78
  Month 42 | -1.6 (5.1) | -0.9 (4.1) | -2.3 (4.0)
  Month 48: number analyzed (Participants) | 254 | 438 | 60
  Month 48 | -1.1 (4.8) | -0.8 (3.9) | -1.9 (4.0)
  Month 54: number analyzed (Participants) | 238 | 387 | 49
  Month 54 | -1.7 (4.8) | -0.8 (4.1) | -1.2 (4.4)
  Month 60: number analyzed (Participants) | 213 | 324 | 52
  Month 60 | -2.0 (4.9) | -0.6 (4.0) | -1.0 (5.3)
  Month 66: number analyzed (Participants) | 183 | 317 | 38
  Month 66 | -1.1 (4.5) | -0.8 (4.0) | -2.4 (4.6)
  Month 72: number analyzed (Participants) | 150 | 293 | 36
  Month 72 | -1.9 (4.8) | -0.6 (3.7) | -1.6 (3.2)
  Month 78: number analyzed (Participants) | 143 | 247 | 32
  Month 78 | -1.5 (4.7) | -0.6 (4.5) | -1.7 (4.2)
  Month 84: number analyzed (Participants) | 96 | 201 | 25
  Month 84 | -2.3 (4.9) | -0.8 (4.5) | -1.2 (4.5)
  Month 90: number analyzed (Participants) | 93 | 176 | 21
  Month 90 | -1.9 (4.7) | -0.9 (3.9) | -2.0 (3.9)
  Month 96: number analyzed (Participants) | 78 | 164 | 19
  Month 96 | -2.4 (4.3) | -1.0 (3.8) | -1.6 (4.2)
  Month 102: number analyzed (Participants) | 28 | 49 | 12
  Month 102 | -1.9 (3.9) | -1.6 (3.9) | -0.3 (3.0)
  Month 108: number analyzed (Participants) | 5 | 14 | 6
  Month 108 | -1.8 (1.9) | -0.8 (5.3) | 0.0 (1.5)

4. Secondary Outcome: Change From Baseline in Patient's Harvey Bradshaw Index (HBI) Total Score to Each Post-Baseline Assessment
Description: HBI response determined based on patient reported HBI total scores was defined as a drop of at least 3 points from baseline HBI total score. Patient reported HBI was composed of 4 parameters: the general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), and whether there are any complications [1 per item: joint pain (arthralgia), eye inflammation (uveitis), red nodules on skin (erythema nodosum), canker sores (aphthous ulcers), skin wound/ulcers (pyoderma gangrenosum), tear in skin of anal area (anal fissure), fluid or pus drainage from anal area (new fistula), and abscess]. The total HBI score was sum of all the 4 individual parameters, where minimum score was 0 and there was no pre-specified maximum score as it was dependent on the number of liquids stools. Higher HBI scores indicated greater disease activity. A negative change indicated less disease activity.
Time Frame: Month 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81, 84, 87, 90, 93, 96, 99, 102, 105 and 108, compared to Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline)
Number analyzed (Participants) | 1131 | 1666 | 275
units on a scale
  Month 3: number analyzed (Participants) | 632 | 960 | 152
  Month 3 | 0.6 (4.4) | 0.2 (3.5) | 0.1 (4.7)
  Month 6: number analyzed (Participants) | 535 | 801 | 108
  Month 6 | 0.2 (4.9) | -0.1 (3.8) | -0.0 (4.0)
  Month 9: number analyzed (Participants) | 546 | 849 | 115
  Month 9 | -0.0 (4.7) | 0.1 (3.9) | -0.1 (4.7)
  Month 12: number analyzed (Participants) | 532 | 875 | 109
  Month 12 | -0.5 (4.4) | -0.0 (3.8) | 0.1 (4.6)
  Month 15: number analyzed (Participants) | 481 | 817 | 100
  Month 15 | -0.6 (4.4) | -0.2 (3.6) | -0.5 (4.1)
  Month 18: number analyzed (Participants) | 505 | 791 | 100
  Month 18 | -0.7 (4.6) | -0.1 (3.6) | -0.3 (4.0)
  Month 21: number analyzed (Participants) | 491 | 801 | 97
  Month 21 | -0.7 (4.9) | -0.2 (3.6) | 0.3 (5.5)
  Month 24: number analyzed (Participants) | 510 | 820 | 112
  Month 24 | -0.6 (5.1) | -0.1 (3.6) | -0.8 (4.7)
  Month 27: number analyzed (Participants) | 475 | 780 | 103
  Month 27 | -0.6 (4.9) | -0.0 (3.6) | -0.1 (4.7)
  Month 30: number analyzed (Participants) | 459 | 779 | 105
  Month 30 | -0.7 (5.0) | -0.1 (3.7) | -0.3 (5.3)
  Month 33: number analyzed (Participants) | 449 | 756 | 102
  Month 33 | -0.9 (4.8) | -0.1 (3.7) | -0.3 (5.0)
  Month 36: number analyzed (Participants) | 439 | 746 | 95
  Month 36 | -0.6 (5.6) | -0.3 (4.0) | -0.6 (6.0)
  Month 39: number analyzed (Participants) | 415 | 714 | 92
  Month 39 | -0.5 (5.8) | -0.3 (3.6) | -0.8 (5.3)
  Month 42: number analyzed (Participants) | 395 | 685 | 89
  Month 42 | -0.4 (4.8) | -0.2 (3.9) | -0.8 (5.2)
  Month 45: number analyzed (Participants) | 393 | 662 | 83
  Month 45 | -0.5 (4.7) | -0.0 (4.1) | -1.2 (4.4)
  Month 48: number analyzed (Participants) | 375 | 652 | 76
  Month 48 | -0.7 (5.1) | -0.0 (4.0) | -0.1 (4.7)
  Month 51: number analyzed (Participants) | 360 | 617 | 70
  Month 51 | -0.5 (5.0) | -0.1 (4.3) | -0.8 (5.0)
  Month 54: number analyzed (Participants) | 351 | 580 | 66
  Month 54 | -0.6 (4.9) | -0.2 (4.0) | -0.6 (7.7)
  Month 57: number analyzed (Participants) | 330 | 570 | 69
  Month 57 | -1.0 (4.9) | -0.2 (3.8) | -1.1 (5.9)
  Month 60: number analyzed (Participants) | 328 | 537 | 63
  Month 60 | -1.2 (4.8) | -0.2 (4.3) | -0.6 (6.2)
  Month 63: number analyzed (Participants) | 303 | 528 | 63
  Month 63 | -1.2 (4.6) | -0.4 (3.8) | -0.3 (5.7)
  Month 66: number analyzed (Participants) | 282 | 513 | 65
  Month 66 | -1.1 (4.9) | -0.2 (4.0) | -0.2 (6.7)
  Month 69: number analyzed (Participants) | 279 | 476 | 59
  Month 69 | -1.0 (4.7) | -0.3 (3.8) | -0.7 (5.3)
  Month 72: number analyzed (Participants) | 260 | 453 | 49
  Month 72 | -0.8 (5.1) | -0.2 (3.9) | -1.0 (3.9)
  Month 75: number analyzed (Participants) | 243 | 420 | 45
  Month 75 | -0.6 (5.9) | -0.1 (4.7) | -1.1 (3.6)
  Month 78: number analyzed (Participants) | 236 | 415 | 47
  Month 78 | -1.0 (5.1) | -0.1 (4.1) | -0.6 (4.7)
  Month 81: number analyzed (Participants) | 214 | 383 | 46
  Month 81 | -1.1 (5.1) | -0.3 (4.0) | -0.5 (3.2)
  Month 84: number analyzed (Participants) | 193 | 369 | 44
  Month 84 | -1.0 (5.0) | -0.3 (4.2) | -0.5 (3.0)
  Month 87: number analyzed (Participants) | 193 | 333 | 36
  Month 87 | -0.5 (5.4) | -0.2 (4.4) | -0.5 (3.5)
  Month 90: number analyzed (Participants) | 168 | 299 | 33
  Month 90 | -0.7 (5.2) | 0.0 (4.7) | 0.3 (5.2)
  Month 93: number analyzed (Participants) | 158 | 287 | 33
  Month 93 | -1.3 (5.0) | -0.4 (4.3) | -0.6 (3.4)
  Month 96: number analyzed (Participants) | 122 | 232 | 34
  Month 96 | -1.1 (5.7) | -0.5 (4.6) | 0.3 (3.3)
  Month 99: number analyzed (Participants) | 27 | 57 | 19
  Month 99 | -2.2 (6.1) | -0.4 (3.9) | -0.6 (3.5)
  Month 102: number analyzed (Participants) | 9 | 9 | 7
  Month 102 | 0.2 (3.3) | 0.2 (2.4) | 1.3 (3.7)
  Month 105: number analyzed (Participants) | 2 | 3 | 6
  Month 105 | -1.5 (2.1) | 2.3 (2.3) | 0.7 (2.6)
  Month 108: number analyzed (Participants) | 1 | 3 | 7
  Month 108 | 8.0 | 2.0 (1.7) | 1.3 (3.0)

5. Secondary Outcome: Change From Baseline in Physician's Assessment of Disease Total Score to Each Post-Baseline Assessment
Description: Physician assessment of disease severity was measured by the general well-being component of HBI score and had a score range of 0= very well to 4= terrible. Higher scores indicated greater disease activity. A negative change indicated less disease activity.
Time Frame: Month 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90, 96, 102, and 108, compared to Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline)
Number analyzed (Participants) | 1131 | 1666 | 275
units on a scale
  Month 6: number analyzed (Participants) | 854 | 1178 | 167
  Month 6 | -0.4 (0.9) | -0.2 (0.8) | -0.3 (0.9)
  Month 12: number analyzed (Participants) | 703 | 1049 | 146
  Month 12 | -0.5 (1.0) | -0.3 (0.9) | -0.3 (0.9)
  Month 18: number analyzed (Participants) | 599 | 954 | 129
  Month 18 | -0.5 (1.0) | -0.3 (0.9) | -0.3 (0.9)
  Month 24: number analyzed (Participants) | 535 | 882 | 121
  Month 24 | -0.6 (1.0) | -0.3 (0.9) | -0.4 (0.9)
  Month 30: number analyzed (Participants) | 458 | 784 | 108
  Month 30 | -0.6 (1.0) | -0.3 (0.9) | -0.4 (0.9)
  Month 36: number analyzed (Participants) | 421 | 698 | 101
  Month 36 | -0.6 (1.0) | -0.4 (0.9) | -0.5 (0.9)
  Month 42: number analyzed (Participants) | 376 | 634 | 94
  Month 42 | -0.6 (1.0) | -0.3 (0.9) | -0.5 (0.8)
  Month 48: number analyzed (Participants) | 334 | 568 | 77
  Month 48 | -0.6 (1.0) | -0.3 (0.9) | -0.4 (0.9)
  Month 54: number analyzed (Participants) | 302 | 496 | 63
  Month 54 | -0.6 (1.0) | -0.4 (1.0) | -0.4 (1.0)
  Month 60: number analyzed (Participants) | 280 | 433 | 64
  Month 60 | -0.7 (1.0) | -0.3 (0.9) | -0.4 (0.9)
  Month 66: number analyzed (Participants) | 244 | 422 | 50
  Month 66 | -0.7 (0.9) | -0.3 (0.9) | -0.4 (0.8)
  Month 72: number analyzed (Participants) | 206 | 376 | 44
  Month 72 | -0.7 (1.0) | -0.3 (1.0) | -0.4 (0.9)
  Month 78: number analyzed (Participants) | 180 | 325 | 42
  Month 78 | -0.7 (0.9) | -0.4 (0.9) | -0.5 (0.9)
  Month 84: number analyzed (Participants) | 124 | 266 | 35
  Month 84 | -0.5 (1.0) | -0.4 (0.9) | -0.5 (0.8)
  Month 90: number analyzed (Participants) | 121 | 224 | 30
  Month 90 | -0.6 (0.9) | -0.4 (0.9) | -0.7 (0.8)
  Month 96: number analyzed (Participants) | 97 | 215 | 26
  Month 96 | -0.6 (1.0) | -0.3 (0.9) | -0.4 (1.0)
  Month 102: number analyzed (Participants) | 34 | 57 | 14
  Month 102 | -0.4 (1.1) | -0.4 (1.1) | -0.1 (0.8)
  Month 108: number analyzed (Participants) | 6 | 16 | 6
  Month 108 | -0.3 (1.0) | -0.1 (1.1) | -0.3 (0.5)

6. Secondary Outcome: Change From Baseline in Patient's Assessment of Disease Total Score to Each Post-Baseline Assessment
Description: Patient assessment of disease severity was measured by the general well-being component of HBI score and had a score range of 0= very well to 4= terrible. Higher scores indicated greater disease activity. A negative change indicated less disease activity.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia at Baseline | No Cimzia at Baseline | Gap (No Cimzia and no Comparator at Baseline)
Number analyzed (Participants) | 1131 | 1666 | 275
units on a scale
  Month 3: number analyzed (Participants) | 636 | 963 | 154
  Month 3 | -0.0 (0.8) | -0.0 (0.7) | -0.1 (0.9)
  Month 6: number analyzed (Participants) | 538 | 803 | 108
  Month 6 | -0.2 (0.9) | -0.1 (0.8) | -0.1 (0.8)
  Month 9: number analyzed (Participants) | 548 | 850 | 115
  Month 9 | -0.2 (0.9) | -0.1 (0.9) | -0.3 (0.9)
  Month 12: number analyzed (Participants) | 534 | 876 | 109
  Month 12 | -0.2 (0.9) | -0.1 (0.8) | -0.2 (0.8)
  Month 15: number analyzed (Participants) | 484 | 819 | 100
  Month 15 | -0.3 (0.9) | -0.1 (0.8) | -0.2 (0.9)
  Month 18: number analyzed (Participants) | 507 | 793 | 100
  Month 18 | -0.3 (0.9) | -0.2 (0.9) | -0.2 (0.8)
  Month 21: number analyzed (Participants) | 494 | 803 | 97
  Month 21 | -0.3 (0.9) | -0.2 (0.8) | -0.3 (1.0)
  Month 24: number analyzed (Participants) | 513 | 822 | 112
  Month 24 | -0.3 (1.0) | -0.2 (0.9) | -0.3 (1.0)
  Month 27: number analyzed (Participants) | 477 | 782 | 103
  Month 27 | -0.3 (1.0) | -0.2 (0.8) | -0.4 (0.9)
  Month 30: number analyzed (Participants) | 461 | 780 | 105
  Month 30 | -0.3 (1.0) | -0.2 (0.8) | -0.4 (0.9)
  Month 33: number analyzed (Participants) | 452 | 759 | 102
  Month 33 | -0.4 (1.0) | -0.2 (0.9) | -0.3 (0.9)
  Month 36: number analyzed (Participants) | 442 | 753 | 95
  Month 36 | -0.4 (1.0) | -0.2 (0.9) | -0.4 (0.9)
  Month 39: number analyzed (Participants) | 418 | 717 | 92
  Month 39 | -0.3 (1.0) | -0.2 (0.9) | -0.3 (1.1)
  Month 42: number analyzed (Participants) | 398 | 686 | 89
  Month 42 | -0.4 (1.0) | -0.2 (0.9) | -0.4 (0.9)
  Month 45: number analyzed (Participants) | 394 | 665 | 83
  Month 45 | -0.3 (1.0) | -0.1 (0.8) | -0.6 (0.8)
  Month 48: number analyzed (Participants) | 376 | 654 | 76
  Month 48 | -0.4 (1.0) | -0.2 (0.8) | -0.3 (0.9)
  Month 51: number analyzed (Participants) | 363 | 620 | 70
  Month 51 | -0.4 (1.0) | -0.2 (0.8) | -0.3 (0.9)
  Month 54: number analyzed (Participants) | 353 | 582 | 66
  Month 54 | -0.4 (1.0) | -0.2 (0.9) | -0.2 (1.0)
  Month 57: number analyzed (Participants) | 332 | 572 | 69
  Month 57 | -0.4 (1.0) | -0.2 (0.8) | -0.4 (0.9)
  Month 60: number analyzed (Participants) | 330 | 539 | 63
  Month 60 | -0.5 (1.0) | -0.3 (0.9) | -0.3 (0.9)
  Month 63: number analyzed (Participants) | 305 | 530 | 63
  Month 63 | -0.5 (1.0) | -0.2 (0.9) | -0.1 (1.0)
  Month 66: number analyzed (Participants) | 284 | 515 | 65
  Month 66 | -0.5 (0.9) | -0.2 (0.8) | -0.3 (0.9)
  Month 69: number analyzed (Participants) | 281 | 476 | 59
  Month 69 | -0.5 (1.0) | -0.2 (0.9) | -0.3 (0.9)
  Month 72: number analyzed (Participants) | 261 | 453 | 49
  Month 72 | -0.5 (0.9) | -0.2 (0.9) | -0.4 (0.8)
  Month 75: number analyzed (Participants) | 244 | 421 | 45
  Month 75 | -0.4 (0.9) | -0.2 (0.9) | -0.4 (0.9)
  Month 78: number analyzed (Participants) | 237 | 416 | 47
  Month 78 | -0.4 (0.9) | -0.2 (0.9) | -0.3 (0.9)
  Month 81: number analyzed (Participants) | 216 | 384 | 46
  Month 81 | -0.5 (0.9) | -0.3 (0.9) | -0.2 (0.9)
  Month 84: number analyzed (Participants) | 194 | 370 | 44
  Month 84 | -0.5 (0.9) | -0.3 (0.9) | -0.3 (0.9)
  Month 87: number analyzed (Participants) | 194 | 334 | 36
  Month 87 | -0.4 (0.9) | -0.2 (0.9) | -0.2 (0.8)
  Month 90: number analyzed (Participants) | 169 | 300 | 33
  Month 90 | -0.4 (0.9) | -0.2 (0.9) | -0.3 (0.8)
  Month 93: number analyzed (Participants) | 159 | 288 | 33
  Month 93 | -0.4 (0.9) | -0.2 (0.9) | -0.2 (1.0)
  Month 96: number analyzed (Participants) | 122 | 233 | 34
  Month 96 | -0.5 (0.9) | -0.2 (0.9) | 0.0 (0.9)
  Month 99: number analyzed (Participants) | 27 | 57 | 19
  Month 99 | -0.5 (0.9) | -0.2 (0.8) | 0.1 (0.8)
  Month 102: number analyzed (Participants) | 9 | 9 | 7
  Month 102 | 0.1 (0.9) | 0.2 (0.7) | 0.0 (0.6)
  Month 105: number analyzed (Participants) | 2 | 3 | 6
  Month 105 | 0.5 (0.7) | 0.3 (0.6) | 0.3 (0.5)
  Month 108: number analyzed (Participants) | 1 | 3 | 7
  Month 108 | 1.0 | 0.3 (0.6) | 0.4 (0.5)

ADVERSE EVENTS:
Time Frame: From Baseline up to 10 years
Description: Treatment-Emergent adverse events (TEAEs) were defined as those events which first occurred or increased in relationship to treatment after the first dose of any crohn's disease drug following enrollment. Participants were counted in more than one arm based on the various treatments they actually received and presented based on acute event rules. Based upon planned analysis of acute event rules, TEAEs are reported for Cimzia®, Comparator, Overlap, Gap and Any Cimzia® reporting groups.
Groups:
- Cimzia: Participants (exposure and events) while receiving Cimzia® only including the half-life of Cimzia® without comparator including half-life of comparator. Participants may be included in treatment groups.
- Gap (No Cimzia and no Comparator at Baseline): Participants (exposure and events) neither receiving Cimzia® (including the half-life of Cimzia®) nor receiving comparator (including the half-life).
Arm/Group | Cimzia | Comparator | Overlap | Gap (No Cimzia and no Comparator at Baseline) | Cimzia + Overlap
All-Cause Mortality (participants affected / at risk) | 3/824 | 25/2478 | 6/1165 | 17/1022 | 9/1428
Serious Adverse Events (participants affected / at risk) | 145/824 | 638/2478 | 268/1165 | 152/1022 | 385/1428
Other Adverse Events (participants affected / at risk) | 19/824 | 70/2478 | 30/1165 | 9/1022 | 48/1428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimzia (N=824) | Comparator (N=2478) | Overlap (N=1165) | Gap (No Cimzia and no Comparator at Baseline) (N=1022) | Cimzia + Overlap (N=1428)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micrognathia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Persistent urogenital sinus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 5 (6) | 2 (2) | 1 (1) | 5 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 8 (8) | 1 (1) | 0 (0) | 2 (2)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Anal stenosis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 24 (27) | 192 (276) | 101 (143) | 40 (45) | 123 (170)
Colitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 23 (27) | 93 (123) | 23 (33) | 18 (26) | 45 (60)
Small intestinal stenosis (Gastrointestinal disorders) | 6 (6) | 5 (6) | 1 (1) | 0 (0) | 7 (7)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 4 (4)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 28 (37) | 17 (20) | 4 (4) | 19 (22)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (5) | 0 (0) | 6 (7)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 4 (4)
Fistula of small intestine (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pouchitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 24 (26) | 9 (9) | 5 (5) | 12 (13)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 5 (5)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 15 (15) | 7 (7) | 0 (0) | 8 (8)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Jejunal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 3 (3)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 6 (6) | 2 (2) | 1 (1) | 2 (2)
Adhesion (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Obstruction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Food interaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Chest pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abdominal abscess (Infections and infestations) | 5 (5) | 14 (21) | 11 (11) | 0 (0) | 16 (16)
Anal abscess (Infections and infestations) | 4 (4) | 6 (8) | 1 (1) | 0 (0) | 5 (5)
Gastroenteritis (Infections and infestations) | 2 (3) | 3 (3) | 2 (2) | 2 (2) | 4 (5)
Perirectal abscess (Infections and infestations) | 2 (2) | 9 (10) | 6 (6) | 3 (3) | 8 (8)
Abdominal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Abscess intestinal (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Anal fistula infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal fistula infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium chelonae infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium kansasii infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 8 (9) | 9 (9) | 1 (1) | 11 (11)
Anorectal cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stoma site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 9 (9) | 5 (5) | 5 (5) | 7 (7)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 3 (3)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Pelvic abscess (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
Abscess (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 4 (4)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pathogen resistance (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stoma site abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 24 (25) | 10 (10) | 4 (4) | 12 (12)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 11 (14) | 6 (6) | 4 (4) | 7 (7)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 8 (8) | 4 (5) | 2 (2) | 6 (7)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ureteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 4 (4) | 5 (5) | 0 (0) | 7 (7)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (4)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumocephalus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 3 (3)
Stoma site ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 6 (10) | 0 (0) | 2 (2) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cells stool positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal stoma output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal examination (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Norovirus test positive (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appetite disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (5) | 1 (2)
Electrolyte depletion (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 3 (3)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 4 (4) | 2 (3) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 4 (5)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioimmunoblastic T-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic paroxysmal hemicrania (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Status migrainosus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 21 (24) | 8 (8) | 5 (5) | 14 (14)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alcohol problem (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 15 (16) | 4 (4) | 1 (1) | 7 (7)
Renal failure (Renal and urinary disorders) | 1 (1) | 7 (7) | 1 (1) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 11 (11) | 4 (4) | 1 (1) | 7 (7)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hydrosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 3 (3)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 5 (5) | 1 (1) | 7 (7)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic cutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Victim of homicide (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Explorative laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proctectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Transfusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug detoxification (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileocolectomy (Surgical and medical procedures) | 2 (2) | 7 (7) | 2 (2) | 0 (0) | 4 (4)
Intestinal resection (Surgical and medical procedures) | 2 (2) | 12 (12) | 4 (4) | 1 (1) | 6 (6)
Enterostomy (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intestinal anastomosis (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Intestinal operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shoulder arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Caecum operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Colectomy total (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pouch procedure (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proctocolectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Drug rehabilitation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileectomy (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ileostomy (Surgical and medical procedures) | 1 (1) | 5 (5) | 0 (0) | 4 (4) | 1 (1)
Ileostomy closure (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Small intestinal resection (Surgical and medical procedures) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Small intestine operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Adhesiolysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma closure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 8 (8) | 6 (7) | 0 (0) | 7 (8)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimzia (N=824) | Comparator (N=2478) | Overlap (N=1165) | Gap (No Cimzia and no Comparator at Baseline) (N=1022) | Cimzia + Overlap (N=1428)
Crohn's disease (Gastrointestinal disorders) | 6 (7) | 13 (13) | 11 (12) | 1 (1) | 17 (19)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 13 (16) | 6 (6) | 1 (1) | 11 (12)
Clostridium difficile infection (Infections and infestations) | 3 (4) | 13 (21) | 6 (6) | 1 (1) | 9 (10)
Herpes zoster (Infections and infestations) | 2 (2) | 19 (19) | 5 (5) | 3 (3) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (9) | 5 (5) | 2 (2) | 10 (11)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 13 (13) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT00844285/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT00844285/SAP_001.pdf